CLINICAL TRIAL: NCT02585128
Title: Incidence and Risk Factors of Acute Postoperative Confusion State After Trans-catheter Aortic Valve Implantation (TAVI)
Brief Title: Predictors of Postoperative Delirium After Transcatheter Aortic Valve Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiocentro Ticino (Other)
Responsible Party: Principal Investigator, Tiziano Cassina, Tiziano Cassina, MD, Cardiocentro Ticino
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DELTAVI-CCT-ICU-2015
Record Dates: First submitted 2015-10-01; First posted 2015-10-23 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Delirium
Keywords: Delirium; Transcatheter Aortic Valve Implantation; Elderly
MeSH Terms: conditions — Emergence Delirium; Delirium | interventions — Mental Status and Dementia Tests; 4-amino-4'-hydroxylaminodiphenylsulfone; Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients following TAVI (Other)
  Interventions: Other: Delirium assessment; Other: MMSE (Mini Mental State Examination); Other: Barthel index; Other: HADS (Hospital Anxiety and Depression Scale); Other: MNA-SF (Mini Nutritional Assessment - Short Form); Device: NIRS (Near-Infrared Spectroscopy); Other: CIRS (Cumulative Illness Rating Scale)

INTERVENTIONS:
Other: Delirium assessment — During the first post-procedural five days all patients will be evaluated on a daily basis for delirium occurrence by the CAM (Confusion Assessment Method) or CAM - ICU (Confusion Assessment Method - Intensive Care Unit)
Other: MMSE (Mini Mental State Examination)
Other: Barthel index
Other: HADS (Hospital Anxiety and Depression Scale)
Other: MNA-SF (Mini Nutritional Assessment - Short Form)
Device: NIRS (Near-Infrared Spectroscopy) — Regional cerebral oxygen saturation monitoring during TAVI procedure
Other: CIRS (Cumulative Illness Rating Scale)

SUMMARY:
Patients undergoing transcatheter aortic valve implantation (TAVI) have distinctive characteristics: they are old, frail, with several co-morbidities and take multiple medications. Hemodynamic instability, cerebral embolism, sedation, general anesthesia and hospitalization in intensive care expose those patients to postprocedural delirium.

Acute neurocognitive dysfunctions are associated with adverse outcomes in these population.

The objective of this study is to determine the incidence of delirium and neurocognitive disorders in elderly patients after TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Age 65>years
* Patients undergoing transcatheter aortic valve implantation
* Patients have given informed consent for participation at the study

Exclusion Criteria:

* Patient suffering from delirium (CAM diagnosis) at recruitment
* Inability to understand the national languages
* Emergency procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 201 (Actual)
Dates: Start 2015-09; Primary Completion 2019-05 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium | Day 1-5 after transcatheter aortic valve implantation
  The primary outcome is incidence of delirium. Delirium screening will be carry out using the CAM or CAM-ICU in accordance with local hospital clinical delirium-screening guidelines. The assessment of presence of Delirium will be perform by clinician with CAM in agreement with Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM IV). CAM is standardized method to enable non-psychiatrically trained clinicians to identify delirium and assesses nine features of delirium: (1) acute onset, (2) inattention, (3) disorganized thinking, (4) altered level of consciousness, (5) disorientation, (6) memory impairment, (7) perceptual disturbances, (8) psychomotor agitation or retardation and (9) altered sleep-wake cycle. Delirium is diagnosed when feature 1 and 2 are present and either 3 or 4 are displayed.

SECONDARY OUTCOMES:
Risk factors for postoperative delirium | Baseline, intra-operative and days 1-5 after transcatheter aortic valve implantation
  Association between incidence of delirium and patient vulnerabilities, exposure to noxious or precipitating factors. The risk factors will be divided in pre-procedural, intra-procedural and post-procedural
Onset of delirium | Day 1-5 after transcatheter aortic valve implantation
Complications of delirium | Day 1-5 after transcatheter aortic valve implantation
  Complications delirium related
Type of delirium | Day 1-5 after transcatheter aortic valve implantation
  Delirium classification according to Delirium Motor Subtype Scale (DMSS-4)
Trajectories of neurocognitive function | Changes from baseline up to 5 day and 3-months
  Change of Mini-Mental State Examination (MMSE)
Trajectories of functional abilities | Changes from baseline up to 5 day and 3-months
  Change of Barthel Index (for Activities of Daily Living, ADL)
Mortality | 30-days, 3-months and 1 year
  Postoperative survival

OTHER OUTCOMES:
TAVI complications | Participants will be followed for the first 72-96 hours after TAVI
  Complications according to VARC-2 (Valve Academic Research Consortium -2)

CONTACTS AND LOCATIONS:
Overall Officials: Tiziano Cassina, MD, Principal Investigator — Cardiocentro Ticino
Locations (1):
- Cardiocentro Ticino, Lugano, Canton Ticino, Switzerland